CLINICAL TRIAL: NCT06220916
Title: Systematic Registration and Longitudinal Monitoring of Predisposing Factors and Acute/Emergent Events of Higher Vocational Schools' Students.
Brief Title: The Greek Acute Dance Injuries Registry
Acronym: GrADIR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Michail Elpidoforou, Principal Investigator, National and Kapodistrian University of Athens
Other Study IDs: 285/10.05.2023
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Emergencies
Keywords: Dance; Emergent events; Predisposing risk factors; Dance medicine
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Greek National School of Dance - GNSD: All the GNSD undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School of Maria Grigoriou - Choros: All the Choros undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School Chorochronos: All the Chorochronos undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School of Moragemou: All the Moragemou undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School Aktina: All the Aktina undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School of Maro Marmarinou: All the Maro Marmarinou undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School of Athens Conservatoire: All the Athens Conservatoire undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance
- Higher Vocational Dance School of Marias Chatzimihali Charlafti: All the Marias Chatzimihali Charlafti undergraduate students with written consent for participating into the study
  Interventions: Behavioral: Dance training in Classical Ballet and Contemporary Dance

INTERVENTIONS:
Behavioral: Dance training in Classical Ballet and Contemporary Dance — Classes, Rehearsals, and Performances of classical ballet and contemporary dance.

SUMMARY:
Dance is a highly demanded physical activity with a high rate of acute and emergent events (AEE). No systematic prospective study has been conducted in any Greek population of dance students for the registration of the AEE and their possible predisposing factors. This is a prospective cohort study, the purpose of which is to register the AEE risk factors, their long-term follow-up, and the potential AEE during an academic year in adult dance students in Athens, Greece.

DETAILED DESCRIPTION:
Dance, as a physical activity, is considered as one of the most demanding activities at a young age with a high rate of acute and emergent events (AEE). Although dancers perform movement combinations that require high athletic ability, often their physical fitness levels appear to be unexpectedly low and the majority of them will experience at least one injury a year. Determination of the AEE predisposing factors in dancers is necessary to reduce their percentage rates, and until now no systematic prospective study has been conducted in a Greek population of vocational dance schools' students to register both the AEE themselves and their possible predisposing factors.

The primary objective of the study is to register the risk factors for the AEE occurrence in students at Higher Vocational Schools of Dance in Athens and their long-term follow-up. Secondary objectives are to register potential AEE during an academic year and to investigate possible correlations of the above parameters, both among themselves and with socio-demographic, anthropometric, psychometric and medical characteristics of the sample. Finally, a translation and cross-cultural adaptation to a Greek population of the Dance Functional Outcome Survey (DFOS) scale will be carried out.

This is a prospective cohort study with the study population being adult students of 8 Higher Vocational Schools of Dance in Athens. A registration of socio-demographic, anthropometric and medical characteristics, as well as an electrocardiogram, will be carried out at the beginning of the academic year. Core stabilization, balance, body composition, aerobic capacity, dance motor control, dance functional ability, quality of life, fatigue, depressive symptoms, anxiety, stress, performance satisfaction, risk for developing eating disorders, athletic burnout, and predisposition to psychological flow will be registered at the beginning and at the end of the academic year.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student in one of the eight Higher Vocational Dance Schools of the study
* Age ≥18 years
* Ability to understand, write and speak Greek
* Written consent for participating into the study

Exclusion Criteria:

* Student listener who is not officially participating to the whole educational program
* Pregnancy
* Deny to participate and/or give a written consent for participating into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the undergraduate students of the eight higher vocational dance schools in Athens-Greece, that participate in the study, they are going to be informed that they could be indorsed in the study according to the aforementioned inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Registration of Possible Acute/Emergent Events (AEE) | Weekly during one 8-month academic year.
  Undergraduate dance students will be asked to report any of their AEE (prevalence and body region), including any acute and/or emergent dysfunction of a tissue/organ which will be lead to at least one day off from any dance activity, and the AEE mechanism during all the weeks of the academic year.
Acute/Emergent Events (AEE) Incidence Rates | AEE incidence rates will be calculated over the 8-month prospective follow-up.
  AEE incidence rates will be calculated per 1000 dance exposures (dance classes, rehearsals, and performances), according to past research [(number of AEE/dance exposures)*1000] (Dang et al, 2020).

SECONDARY OUTCOMES:
Prevalence of Anatomical Variations (AV) | Baseline
  All the participants will be assessed by a registered physiotherapist either positively (incidence of the AV) or negatively (non-incidence of the AV) for the following AV: knee valgus, knee varum, hallux valgus, splay foot, forefoot adduction, hindfoot varum, hindfoot valgus, longitudinal arch cavus, longitudinal arch planus, forward head, cervical lordosis, thoracic kyphosis, scoliosis, lumbar lordosis, and knee hyperextension, according to past publications (Gamboa et al, 2008; Steinberg et al, 2012).
Registration of subscales score of Medical Outcome Study 36-Item Short-Form Health Survey (SF-36) | Baseline, after 8 weeks, and over the 8-month prospective follow-up.
  SF-36 is used to assess Quality of Life (QoL) and consists of eight physical and mental health domains: Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Subscales evaluate health between 0 and 100, and 0 indicates "bad health", 100 indicates "good health". It will be used to assess QoL and to study construct validity of the DFOS-Gr, similar to that tested in the english (Bronner and Urbano, 2018), spanish (de-la-Cruz-Torres et al, 2020), and italian (Contri et al, 2021) version.
Beighton hypermobility score | Baseline
  Beighton-score is 9 point score for the assessment of hypermobility. It investigates the presence of hyperlaxity (yes = 1, no = 0) at both wrists, the fifth metacarpo-phalangeal joints, elbows, knee joints, and the lumbosacral joints. Sum of the items ranges from 0 to 9 points, with higher scores indicating greater joint laxity.
Thomas Test (TT) | Baseline
  TT (also known as Iliacus Test or Iliopsoas Test) is used to measure hip flexors (iliopsoas muscle group, rectus femoris, pectineus, gracillis, tensor fascia latae, and sartorius) flexibility. Participants will be assessed by a registered physiotherapist either positively (non-flexible hip flexors) or negatively (flexible hip flexors) from supine position on the examination table. Participant holds one knee flexed on his/her chest and lowers the tested limb toward the table. Test is positive when the tested hip joint is flexed, and negative when is hyperextended with the tested limb's thigh under the table.
Active Straight Leg Raise (SLR) | Baseline
  SLR is used to measure hamstring (semimembranosus, semitendinosus and biceps femoris) flexibility. Participants will be assessed by a registered physiotherapist either positively (non-flexible hip flexors) or negatively (flexible hip flexors) from supine position on the examination table. Participant actively flexes his tested hip joint with the knee extended and the non-tested limb totally extended on the table. Test is positive when the tested hip joint is flexed more than 90 degrees, and negative when it is flexed less than 90 degrees.
Ober Test (OT) | Baseline
  OT is used to measure tensor fascia latae (TFL) flexibility. Participants will be assessed by a registered physiotherapist either positively (non-flexible TFL) or negatively (flexible TFL) from lateral decubitus position. The evaluator flexes the knee of the tested limb at 90 degrees and abducts and extends the hip until it is level with the trunk. Only gravity then acts to the tested hip joint bringing it on the maximum possible passive adduction. Test is positive when tested limp's knee is off the table, and negative when it is on the table.
Electrocardiogram (ECG) | Baseline
  For the registration of the prevalence of possible cardiac clinical signs, an ECG will be executed and clinically interpreted by a registered cardiologist.
Dance-related Flexibility Assessment | Baseline
  Five assessments with a goniometer in both sides will be executed, according to past research (Yin et al, 2019): passive range of dorsiflexion from supine position, passive range of hip external and internal rotation from prone position, passive range of hip horizontal abduction from supine position, and active range of hip external rotation from standing position (first feet ballet position), with higher ranges of motion indicating greater flexibility.
Prone Plank Test | Baseline and over the 8-month prospective follow-up.
  The participant is asked to lie facing down and rise on their elbows and toes while keeping the body in a straight line. The total time is recorded for the assessment of the core region muscles strength and endurance (more often called as "core stability"). The time is stopped if the participant lowers or lifts his/her body.
Side Plank Test | Baseline and over the 8-month prospective follow-up.
  The participant is asked to lie on his/her side on the elbow with the lower limbs in full extension. Participant is asked to lift the lower limbs so that the hips and back are aligned and mentain this position. The total time is recorded for both sides, right and left, for the assessment of the lateral trunk flexor muscles strength and endurance (more often called as "lateral core stability"). The time is stopped if the participant lowers or lifts his/her pelvis.
Stork Balance Stand Test | Baseline and over the 8-month prospective follow-up.
  The participant is asked to stand on one foot while he/she raises the other foot off the floor. The total time is recorded for both sides, right and left, for the assessment of static balance. The time is stopped if the supported foot is moved away from the starting position and/or the non-supported foot touches the floor. Rahman's et al (2017) categorization will be used: great (>50''), good (40''-50''), typical (25''-39''), acceptable (10''-24''), and poor (<10'') balance.
Bioelectrical Impedance (BI) assessment | Baseline and over the 8-month prospective follow-up.
  BI will be used to assess body mass (kg), body mass index - BMI (kg/cm^2), fat mass (percentage), and muscle mass (kg).
Accelerated Step Test (AST) | Baseline and over the 8-month prospective follow-up.
  AST is a variation of Kasch Step Test for the aerobic capacity evaluation. Participant is asked to step up and down on a 0,305 meter step for 3 minutes following an audible metronome adjusted in 112 beats*min^-1. Resting heart rate (RHR) before the test and Heart Rate Recovery (HRR) one minute after the test finish will be assessed. HRR score closer to RHR score indicates greater aerobic capacity, according to Darr et al (1988).
Dance Technique Screening Instrument (DTSI) | Baseline and over the 8-month prospective follow-up.
  DTSI is a dance-specific motor control instrument, which assesses the dancer's motor control for different body regions during the execution of 3 dance movements: grand plié à la seconde [pelvis, hips, knees, and feet (0-4 points)], dèveloppé à la seconde [pelvis, turn-out, hips, knees, feet (0-5 points), and sautés au premier position [pelvis, hips, knees, feet (0-4 points)]. One point is added for each incorrect body region's execution. A total score from 9 to 13 points indicates a poor technique, from 5 to 8 points indicates a moderate technique, and from 0 to 4 points indicates a good technique.
Dance Functional Outcome Survey (DFOS) | Baseline, after 8 weeks, and over the 8-month prospective follow-up.
  DFOS is a 14-item lower extremity and low back likert-scale questionnaire, which assesses dancer's ability to accomplish activities of daily living (ADL) and dance-specific movements. It has 2 subscales; the first consists of six items regarding ADL and scored with a total of 40 points, and the second consists of eight items regarding technique and scored with a total of 50 points. The DFOS-total is both sections combined, for a possible score of 90 points, and it is multiplied by 100 to be normalized to a percentage (Bronner et al, 2019).
Multidimensional Fatigue Inventory (MFI) | Baseline and over the 8-month prospective follow-up.
  MFI is a 20-item instrument to measure five dimensions of fatigue (general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue), each item is scored from one to five and each dimension consists of five items. The dimensional score consequently ranges from 4 to 20 (a higher score indicates more fatigue).
Depression Score in Depression, Anxiety and Stress Scale 21 (DASS-21) | Baseline and over the 8-month prospective follow-up.
  Normal score: 0-9, Mild score: 10-12, Moderate score: 13-20, Severe score: 21-27, and Extremely severe: 28-42.
Anxiety Score in Depression, Anxiety and Stress Scale 21 (DASS-21) | Baseline and over the 8-month prospective follow-up.
  Normal score: 0-6, Mild score: 7-9, Moderate score: 10-14, Severe score: 15-19, and Extremely severe: 20-42.
Stress Score in Depression, Anxiety and Stress Scale 21 (DASS-21) | Baseline and over the 8-month prospective follow-up.
  Normal score: 0-10, Mild score: 11-18, Moderate score: 19-26, Severe score: 27-34, and Extremely severe: 35-42.
Performance Satisfaction Scale (PSS) | Baseline and over the 8-month prospective follow-up.
  PSS is a 1-item likert-scale questionnaire to assess the level of dance performance satisfaction, as it is used in past studies (Dotti et al, 1998; Yannakoulia et al, 2004). Total score ranges from 1 (i am not satisfied at all) to 10 (i am absolutely satisfied).
Eating Attitudes Test (EAT-26) | Baseline and over the 8-month prospective follow-up.
  The EAT-26 is a 26-item scale. Items are presented in a 6-point Likert-scale ranging from 1 ("never") to 6 ("always). The total score is obtained re-coding scores as follows: scores from 1 to 3 are re-coded as 0, 4 is re-coded as 1, 5 as 2, and 6 is recoded as 3. The only exception is item 25 whose answers score as follows: 1 as 3, 2 as 2, 3 as 1, and 4 to 6 as 0. The EAT-26 total score ranges from 0 to 78. A higher score indicates greater levels of attitudes and behaviors related to eating disorders.
Athlete Burnout Questionnaire (ABQ) | Baseline and over the 8-month prospective follow-up.
  Greek version of ABQ is a 13-item scale that evaluates the 3 constructs of athlete burnout: emotional or physical exhaustion, reduced sense of accomplishment, and sport devaluation. Each item is rated on a 5-point Likert scale ranging from almost never (1) to almost always (5). To calculate average scores for each construct of athlete burnout, subscale scores were summed individually and divided by 5. Higher scores indicate higher burnout levels.
Dispositional Flow Scale-2 (DFS-2) | Baseline and over the 8-month prospective follow-up.
  DFS-2 is a 36-item scale of a 5-point Likert-scale questionnaire ranges from 1 (totally disagree) to 5 (totally agree), with four items for each one of the following nine components (also known as factors and dimensions): Challenge-Skill Balance (CSB), Merging of Action-Awareness (MAA), Clear Goals (CG), Unambiguous Feedback (UF), Concentration on Task at Hand (CTH), Sense of Control (SC), Loss of Self-Consciousness (LSC), Transformation of Time (TT), and Autotelic Experience (AE).

CONTACTS AND LOCATIONS:
Overall Officials: Michail Elpidoforou, MSc, Principal Investigator — Department of Emergency Medicine, Attikon University Hospital
Locations (1):
- Michail Elpidoforou, Chaïdári, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Contri A, Breda G, Vanti C, Pillastrini P, Bronner S. The Dance Functional Outcome Survey: Cultural Adaptation and Psychometric Validation in Italian (DFOS-IT). Med Probl Perform Art. 2021 Sep;36(3):150-162. doi: 10.21091/mppa.2021.3018. PMID 34464961
- [Background] Bronner S, Chodock E, Urbano IER, Smith T. Psychometric Properties of the Dance Functional Outcome Survey (DFOS): Reliability, Validity, and Responsiveness. J Orthop Sports Phys Ther. 2019 Feb;49(2):64-79. doi: 10.2519/jospt.2019.8247. Epub 2018 Jul 27. PMID 30053790
- [Background] Bronner S, Urbano IR. Dance Functional Outcome Survey: Development and Preliminary Analyses. Sports Med Int Open. 2018 Nov 28;2(6):E191-E199. doi: 10.1055/a-0729-3000. eCollection 2018 Nov. PMID 30539138
- [Background] de-la-Cruz-Torres B, Barrera-Garcia-Martin I, Romero-Morales C, Bronner S. Cross-Cultural Adaptation of the Dance Functional Outcome Survey (DFOS) for Spanish Dancers. Diagnostics (Basel). 2020 Mar 20;10(3):169. doi: 10.3390/diagnostics10030169. PMID 32245063
- [Background] Dotti A, Lazzari R. Validation and reliability of the Italian EAT-26. Eat Weight Disord. 1998 Dec;3(4):188-94. doi: 10.1007/BF03340009. PMID 10728170
- [Background] Yannakoulia M, Matalas AL, Yiannakouris N, Papoutsakis C, Passos M, Klimis-Zacas D. Disordered eating attitudes: an emerging health problem among Mediterranean adolescents. Eat Weight Disord. 2004 Jun;9(2):126-33. doi: 10.1007/BF03325056. PMID 15330080
- [Background] Dang Y, Koutedakis Y, Wyon M. Fit to Dance Survey: Elements of Lifestyle and Injury Incidence in Chinese Dancers. Med Probl Perform Art. 2020 Mar;35(1):10-18. doi: 10.21091/mppa.2020.1002. PMID 32135000
- [Background] Gamboa JM, Roberts LA, Maring J, Fergus A. Injury patterns in elite preprofessional ballet dancers and the utility of screening programs to identify risk characteristics. J Orthop Sports Phys Ther. 2008 Mar;38(3):126-36. doi: 10.2519/jospt.2008.2390. PMID 18383646
- [Background] Steinberg N, Siev-Ner I, Peleg S, Dar G, Masharawi Y, Zeev A, Hershkovitz I. Extrinsic and intrinsic risk factors associated with injuries in young dancers aged 8-16 years. J Sports Sci. 2012;30(5):485-95. doi: 10.1080/02640414.2011.647705. Epub 2012 Jan 30. PMID 22288886
- [Background] Yin AX, Geminiani E, Quinn B, Owen M, Kinney S, McCrystal T, Stracciolini A. The Evaluation of Strength, Flexibility, and Functional Performance in the Adolescent Ballet Dancer During Intensive Dance Training. PM R. 2019 Jul;11(7):722-730. doi: 10.1002/pmrj.12011. Epub 2019 Feb 13. PMID 30758918
- [Background] Darr KC, Bassett DR, Morgan BJ, Thomas DP. Effects of age and training status on heart rate recovery after peak exercise. Am J Physiol. 1988 Feb;254(2 Pt 2):H340-3. doi: 10.1152/ajpheart.1988.254.2.H340. PMID 3344824